CLINICAL TRIAL: NCT04765410
Title: Tissue Micro-RNA Profile Collected Through Endoscopic Ultrasonography Fine-Needle-Aspiration (EUS-FNA) In Pancreatic Adenocarcinoma And Its Impact On Survival And Prognosis
Brief Title: The Impact Of Tissue Micro-RNA Profile From EUS-FNA In Pancreatic Adenocarcinoma
Acronym: EUS-FNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Carol Davila University of Medicine and Pharmacy (Other)
Collaborators: Bucharest Emergency Hospital (Other); Institutul Clinic Fundeni (Other)
Responsible Party: Principal Investigator, Mihai Ciocirlan, MD PhD, Carol Davila University of Medicine and Pharmacy
Other Study IDs: PDACmiRNA
Record Dates: First submitted 2021-02-18; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: microRNA; endoscopic ultrasonography; fine needle aspiration
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The samples will be obtained from the participants during endoscopic ultrasonography, through fine needle aspiration, after consent was given to be a part of the study prior to the intervention. The probe will be preserved in a special recipient that stabilizes RNA and inhibits RNA-lazes, thus preventing RNA degradation by endogenous ribonucleases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with solid pancreatic masses: Patients with solid pancreatic masses
  Interventions: Diagnostic Test: EUS FNA (endoscopic ultrasound fine needle aspiration)

INTERVENTIONS:
Diagnostic Test: EUS FNA (endoscopic ultrasound fine needle aspiration) — Patients with solid pancreatic masses fulfilling the inclusion and exclusion criteria will receive EUS FNA (endoscopic ultrasound fine needle aspiration).

SUMMARY:
Pancreatic adenocarcinoma still represents one of the "hot-topics" worldwide. Endoscopic ultrasonography was a breakthrough, bringing us closer to personalized treatment by getting histopathological samples through fine-needle-aspiration or fine-needle-biopsy. These samples can be analyzed and offer the possibility to detect a micro-RNA profile.

Micro-RNAs are small non-coding RNA molecules that interfere in genic expression. Many studies focused on seric microRNA profile, though there are many implications in tissue micro-RNA profile, thus overexpression or under expression of these molecules might help us not only understand different cellular processes, but also interfere in personalized medicine in the future.

The investigators propose a prospective, multicenter, randomized, cohort study on 60 patients with solid pancreatic masses to evaluate tissue microRNA profile obtained by EUS-FNA.

The primary hypothesis is to correlate the microRNA tissular expression in pancreatic adenocarcinoma with tumor aggressive behavior, survival and response to treatment.

The samples will be obtained from the participants during endoscopic ultrasonography, through fine needle aspiration, after consent was given to be a part of the study prior to the intervention. The probe will be preserved in a special recipient that stabilizes RNA and inhibits RNA-lazes, thus preventing RNA degradation by endogenous ribonucleases.

The analysis of miRNA profile will be made using qRT-PCR array method, by miScript II RT Kit, miScript SYBR Green PCR Kit și miScript miRNA PCR Array Human Cancer Pathway Finder (MIHS-102Z) (Qiagen, GmbH). Thus a kit containing a number of 84 miRNAs will be analysed in every participant.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic solid mass, with or without a cystic component
* Age over 18 years old
* Signed informed consent

Exclusion Criteria:

* Cystic pancreatic mass with no solid component
* Abnormal coagulation (elevated INR >1.5, thrombocytopenia<60 000/mm3, activated partial thromboplastin time>42 seconds), participant on anticoagulant treatment that cannot stop the treatment
* European Cooperative Oncology Group status 4
* Pregnancy
* Age under 18 years old
* The participant does not want to sign the consent form, or is unable to
* Difficult puncture position during endoscopic ultrasonography: vessels or Wirsung duct positioned in front of the needle (decision of the endoscopist)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid pancreatic masses fulfilling the inclusion and exclusion criteria will receive EUS FNA (endoscopic ultrasound fine needle aspiration).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-03-21 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Mean change from baseline in Eastern Cooperative Oncology Group (ECOG) performance status, weight and survival in patients with pancreatic adenocarcinoma according to tissue microRNA expression | through study completion, an average of 2 and a half years
  Eastern Cooperative Oncology Group (ECOG) performance status, weight and survival will be assessed though different consultations (in person or by telemedicine): at first presentation, at 1 month, at 3 months, at 6 months and at one year.

CONTACTS AND LOCATIONS:
Locations (5):
- Romania (5):
  - "Carol Davila" University Central Emergency Hospital, Bucharest, Sector 1
  - "Prof Dr Agrippa Ionescu" Emergency Hospital, Bucharest, Sector 1
  - Clinical Emergency Hospital Bucharest, Bucharest, Sector 1
  - Fundeni Clinical Institute, Bucharest, Sector 2
  - "Victor Babes" National Pathology Institute, Bucharest, Sector

IPD SHARING:
Plan to Share IPD: Undecided